CLINICAL TRIAL: NCT05498857
Title: Intramuscular Ephedrine in the Prevention of Hypotension in Patients Undergoing Spinal Anesthesia: a Prospective, Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Intramuscular Ephedrine in the Prevention of Hypotension in Patients Undergoing Spinal Anesthesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Base (Other)
Responsible Party: Principal Investigator, Fabricio Tavares Mendonca, MD, MSc, PhD, Hospital de Base
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: i.m. ephedrine
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Ephedrine; Intramuscular; Hypotension; Spinal Anesthesia
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blind and placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ephedrine group (Active Comparator): Patients will receive intramuscular ephedrine 0,5 mg/kg before spinal anesthesia
  Interventions: Drug: Intramuscular ephedrine; Drug: Placebo
- Placebo group (Placebo Comparator): Patients will receive intramuscular saline before spinal anesthesia
  Interventions: Drug: Intramuscular ephedrine; Drug: Placebo

INTERVENTIONS:
Drug: Intramuscular ephedrine — Patients will receive prophylactic intramuscular ephedrine plus standard spinal anesthesia
Drug: Placebo — Patients will receive prophylactic intramuscular saline plus standard spinal anesthesia

SUMMARY:
Subarachnoid anesthesia is an alternative and usually the first choice for many surgical procedures. It is a simple and safe procedure, however it can present complications such as hypotension and bradycardia. In this sense, ephedrine, an alpha and beta agonist agent, commonly used as rescue therapy for these events, is also potentially useful for prophylaxis of this unwanted effect and for less hemodynamic variation when preventively administered via the intramuscular route. Two groups will be divided: intramuscular ephedrine (0.5 mg/kg) and placebo. The variables analyzed and compared will be the incidence of hypotension and bradycardia, variation in mean and systolic blood pressure, heart rate, in addition to side effects. The main objective is to verify if the use of intramuscular ephedrine prior to spinal block is able to reduce the incidence of hypotension.

DETAILED DESCRIPTION:
Subarachnoid or spinal anesthesia is an alternative and usually the first choice for many surgical procedures of the lower limbs, perineum and lower abdomen. It is a simple and safe procedure, however it can present complications such as hypotension and bradycardia. The incidence of hypotension and bradycardia is approximately 30 and 10%, respectively, during spinal anesthesia, however, the incidence of hypotension can be as high as 50 to 60% in obstetric patients.

In this sense, it is common for ephedrine, an agent with beta and alpha agonist action, to be the medication of first choice for rescuing hypotension and bradycardia after subarachnoid block, with part of its action happening by a direct mechanism and part by stimulus and indirect release. of endogenous catecholamines stored in the adrenal.

It is known that intramuscular administration has slower absorption and lower bioavailability of the drug compared to intravenous administration. Therefore, we have in our favor: a later serum peak, coinciding with the establishment of sympathetic block after spinal anesthesia, as well as more insidious effects, with less tendency to peaks and valleys and greater hemodynamic stability when compared to therapy alone. intravenous rescue. To assess this response, the main objective of the present study is to verify the hypothesis that the previous administration of ephedrine by intramuscular route reduces the incidence of hypotension induced by spinal anesthesia.

The proposal is a prospective, randomized, double-blind, placebo-controlled study in surgical procedures. Examiners responsible for evaluating patients will not have access to the agents used. Patients will be randomized through a list generated by lottery. The examiner responsible for opening the envelope, will perform the drawing, include the patient in one of the groups, write down his/her data in the random list, prepare the syringe with the medication, and deliver it to the operating room so that the following examiners will not be aware of the administered drug.

Patients will receive standard monitoring, venoclysis, intravenous midazolam as pre-anesthetic medication. Then, the study drug will be administered (ephedrine 0.3mg/kg intramuscularly or placebo). All patients received spinal anesthesia with hyperbaric bupivacaine and opioid adjuvants at the discretion of the anesthesiologist, except clonidine.

The evolution of vital signs such as systolic and mean blood pressure, heart rate, height of sensory block, incidence of adverse events such as bradycardia, tachycardia, hypertension or hypotension, nausea, vomiting, consumption of vasopressors and antiemetics will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old, electively scaled for surgery requiring neuraxial block, with programming of spinal anesthesia.
* Physical State 1, 2 or 3 of the American Society of Anesthesiology (ASA)

Exclusion Criteria:

* Patients taking prophylactic or therapeutic anticoagulation, except respecting the allowed range;
* Patients with atrioventricular block
* Patients with cardiac arrhythmias
* Patients with heart failure;
* Patients with renal disease
* Patients with liver disease
* Patient carrying or suspecting any type of systemic infection or located in a puncture site;
* Patients who refuse to participate in the study after presenting the free and informed consent form;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events as hypotension | During surgery
  Intraoperative hemodynamic stability analysis through the incidence of bradycardia, hypotension and consumed vasopressors

CONTACTS AND LOCATIONS:
Overall Officials: Fabricio T Mendonca, MD, MSc, PhD, Principal Investigator — Hospital de Base do Distrito Federal
Locations (1):
- Hospital de Base do Distrito Federal, Brasília, Federal District, Brazil